CLINICAL TRIAL: NCT01085708
Title: A Pilot Cross-over Bioequivalence Study of E3810 for Healthy Japanese Male (Under Postprandial Condition)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E3810-J081-034
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Rabeprazole; Japan; healthy Japanese male
MeSH Terms: interventions — Rabeprazole

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: rabeprazole
- 2 (Experimental)
  Interventions: Drug: rabeprazole
- 3 (Experimental)
  Interventions: Drug: rabeprazole
- 4 (Active Comparator)
  Interventions: Drug: rabeprazole

INTERVENTIONS:
Drug: rabeprazole — 10 mg normal tablet
  Arms: 1
Drug: rabeprazole — Type 1 granule containing rabeprazole 10 mg
  Arms: 2
Drug: rabeprazole — Type 2 granules containing rabeprazole 10 mg
  Arms: 3
Drug: rabeprazole — Type 3 granules containing rabeprazole 10 mg
  Arms: 4

SUMMARY:
The purpose of this study is to assess pharmacokinetics of rabeprazole under postprandial condition.

ELIGIBILITY:
Inclusion criteria:

Subjects with homozygous or heterozygous extensive metabolizers of cytochrome P4502C19

Exclusion criteria:

Subjects with allergy

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The following pharmacokinetic parameters are calculated: maximum drug concentration (Cmax) in plasma; area under the plasma concentration time curve (AUC) | One day

CONTACTS AND LOCATIONS:
Overall Officials: Kai Shibata, Study Director — Clinical Research Center, Eisai, Co., Ltd